CLINICAL TRIAL: NCT02905214
Title: Coroflex ISAR 2000 Extended Postmarket Surveillance Non-Interventional Study
Brief Title: Coroflex ISAR 2000 Extended Registry (ISAR2000 Extended)
Status: Completed | Type: Observational
Sponsor: B. Braun Melsungen AG (Industry)
Collaborators: Charite University, Berlin, Germany (Other)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1601
Record Dates: First submitted 2016-09-14; First posted 2016-09-19 (Estimated); Last update posted 2022-02-08 (Actual); Status verified 2022-02

CONDITIONS: Coronary Artery Disease (CAD)
MeSH Terms: conditions — Coronary Artery Disease | interventions — Stents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: stenting with the Coroflex ISAR sirolimus-eluting stent — coronary stenting
  Other Names: Coroflex ISAR

SUMMARY:
Postmarket surveillance in terms of the safety and efficacy of Sirolimus-eluting Coroflex ISAR Stent for the treatment of "real world" patients with de-novo and restenotic lesions after stand-alone angioplasty in coronary arteries.

DETAILED DESCRIPTION:
The aim of the study is to assess the safety and efficacy of elective deployment of the Sirolimus-eluting Coroflex ISAR Stent for the treatment of "real world" de-novo and restenotic lesions after stand-alone angioplasty in coronary arteries of 2.0 mm up to 4.0 mm in diameter and up to 30 mm in length for procedural success and preservation of vessel patency.

ELIGIBILITY:
Inclusion Criteria:

* patients suitable for percutaneous coronary intervention with proof of ischemia
* at least 18 years of age

Exclusion Criteria:

* Intolerance to sirolimus and/or probucol
* Allergy to components of the coating
* Pregnancy and lactation
* Complete occlusion of the treatment vessel
* Severely calcified stenosis
* Cardiogenic shock
* Risk of an intraluminal thrombus
* Haemorrhagic diathesis or another disorder such as gastro-intestinal ulceration or cerebral circulatory disorders which restrict the use of platelet aggregation inhibitor therapy and anti-coagulation therapy
* Surgery shortly after myocardial infarction with indications of thrombus or poor coronary flow behavior
* Severe allergy to contrast media
* Lesions which are untreatable with PTCA or other interventional techniques
* Patients with an ejection fraction of < 30 %
* Vascular reference diameter < 2.00 mm
* Treatment of the left stem (first section of the left coronary artery)
* Indication for a bypass surgery
* Contraindication for whichever accompanying medication is necessary

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Unselected patients with coronary de-novo and/or restenotic lesions
Sampling Method: Non-Probability Sample
Enrollment: 4369 (Actual)
Dates: Start 2016-01; Primary Completion 2018-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
clinically driven Target Lesion Revascularization | 9 months
  re-intervention of the target lesion

SECONDARY OUTCOMES:
Major Adverse Cardiac Events | 9 months
  MACE=TLR+MI+cardiac/unknown death
Myocardial infarction rate | 9 months
  myocardial infarction
Cardiac death rate | 9 months
  cardiac death including death of unknown causes
Target lesion revascularization rate | 9 months
  TLR=CABG + Re-PCI
Procedural success | immediately after stent implantation (within the first 30 minutes)
  Success rate to cross and treat the coronary lesion
Stent thrombosis rates | 0-9 months
  acute, subacute and 9-month stent thrombosis rates

CONTACTS AND LOCATIONS:
Overall Officials: Florian Krackhardt, MD, Principal Investigator — Charité Virchow Unversity Hospital
Locations (3):
- Charité University Hospital, Berlin, Germany
- Pusat Perubatan Universiti Malaya, Kuala Lumpur, Malaysia
- Hospital General Universitario de Ciudad Real, Ciudad Real, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Massberg S, Byrne RA, Kastrati A, Schulz S, Pache J, Hausleiter J, Ibrahim T, Fusaro M, Ott I, Schomig A, Laugwitz KL, Mehilli J; Intracoronary Stenting and Angiographic Results: Test Efficacy of Sirolimus- and Probucol-Eluting Versus Zotarolimus- Eluting Stents (ISAR-TEST 5) Investigators. Polymer-free sirolimus- and probucol-eluting versus new generation zotarolimus-eluting stents in coronary artery disease: the Intracoronary Stenting and Angiographic Results: Test Efficacy of Sirolimus- and Probucol-Eluting versus Zotarolimus-eluting Stents (ISAR-TEST 5) trial. Circulation. 2011 Aug 2;124(5):624-32. doi: 10.1161/CIRCULATIONAHA.111.026732. Epub 2011 Jul 18. PMID 21768546
- [Derived] Nuruddin AAB, Ahmad WAW, Waliszewski M, Heang TM, Bang LH, Yusof AKM, Abidin IZ, Zuhdi AS, Krackhardt F. Impact of Coronary Stent Architecture on Clinical Outcomes: Do Minor Changes in Stent Architecture Really Matter? Cardiol Ther. 2021 Jun;10(1):175-187. doi: 10.1007/s40119-020-00204-4. Epub 2020 Dec 4. PMID 33275200
- [Derived] Krackhardt F, Waliszewski MW, Kherad B, Barth C, Marcelli D. Clinical outcomes following polymer-free sirolimus-eluting stent implantations in unselected patients: A descriptive subgroup analysis in patients with renal impairment. Medicine (Baltimore). 2020 Jul 17;99(29):e21244. doi: 10.1097/MD.0000000000021244. PMID 32702903
- [Derived] Krackhardt F, Waliszewski M, Kocka V, Tousek P, Janek B, Hudec M, Lozano F, Roman KG, Del Blanco BG, Mauri J, Heang TM, Ahn TH, Jeong MH, Herberger D, Tomulic V, Levy G, Sebagh L, Rischner J, Pansieri M. Real-World Dual Antiplatelet Therapy Following Polymer-Free Sirolimus-Eluting Stent Implantations to Treat Coronary Artery Disease. Cardiovasc Drugs Ther. 2020 Jun;34(3):335-344. doi: 10.1007/s10557-020-06963-5. PMID 32212061
- [Derived] Krackhardt F, Kocka V, Waliszewski M, Tousek P, Janek B, Trencan M, Krajci P, Lozano F, Roman KG, Otaegui I, Del Blanco BG, Del Olmo VV, Nofrerias EF, Wachowiak L, Heang TM, Ahn TH, Jeong MH, Jung BC, Han KR, Piot C, Sebagh L, Rischner J, Pansieri M, Leschke M. Unrestricted use of polymer-free sirolimus eluting stents in routine clinical practice. Medicine (Baltimore). 2020 Feb;99(8):e19119. doi: 10.1097/MD.0000000000019119. PMID 32080086
- [Derived] Krackhardt F, Waliszewski M, Wan Ahmad WA, Kocka V, Tousek P, Janek B, Trencan M, Krajci P, Lozano F, Garcia-San Roman K, Otaegui Irurueta I, Garcia Del Blanco B, Wachowiak L, Vilalta Del Olmo V, Fernandez Nofrerias E, Ho Jeong M, Jung BC, Han KR, Piot C, Sebagh L, Rischner J, Pansieri M, Leschke M, Ahn TH. Polymer-free sirolimus-eluting stent use in Europe and Asia: Ethnic differences in demographics and clinical outcomes. PLoS One. 2020 Jan 13;15(1):e0226606. doi: 10.1371/journal.pone.0226606. eCollection 2020. PMID 31929543